CLINICAL TRIAL: NCT00754429
Title: The Effect of Losartan Versus Amlodipine-based Antihypertensive Therapy on Atherosclerotic Inflammatory Markers and Cerebrovascular Regulation in Ischemic Stroke Patients
Brief Title: The Effect of Losartan Versus Amlodipine-based Therapy in Ischemic Stroke (0954-338)(COMPLETED)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Executive Vice President, Clinical and Quantitative Sciences, Merck & Co., Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008_025; MK0954-338
Record Dates: First submitted 2008-09-16; First posted 2008-09-18 (Estimated); Last update posted 2013-10-23 (Estimated); Status verified 2013-10

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Losartan; Amlodipine

ARMS (2):
- A (Experimental): Losartan 50mg qd for 30 weeks, if blood pressure > 140/90, or mean arterial Bp ≧ 15% of baseline, then add on diuretics.
  Interventions: Drug: losartan
- B (Active Comparator): Amlodipine 5 mg q.d for 30 weeks, if blood pressure > 140/90, or mean arterial Bp ≧ 15% of baseline, then add on diuretics.
  Interventions: Drug: amlodipine

INTERVENTIONS:
Drug: losartan — losartan 50mg qd for 30 weeks.
  Other Names: losartan potassium; COZAAR®; MK0954
  Arms: A
Drug: amlodipine — amlodipine 5 mg q.d for 30 weeks.
  Other Names: Norvasc
  Arms: B

SUMMARY:
To compare the effect of losartan vs amlodipine-based antihypertensive therapy on atherosclerotic inflammatory markers and cerebrovascular regulation in Ischemic stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient With Tia Or Ischemic Stroke (Event Has Occurred More Thaan 4 Weeks But Less Than 24 Weeks, And Modified Rankin'S Scale, Mrs<=3) With Mild To Moderate Hypertension
* Patient Has No Other Active Medical Problem, Which Might Of Itself Or By This Treatment Significantly Affect The Patient's Blood Pressure
* The Blood Level Of Hscrp>0.2 Ng/Dl By Two Measurements Performed Respectively One-Week Apart

Exclusion Criteria:

* Patients With Cardiac Arrhythmia
* Diabetes Mellitus
* Patient With Other Active Inflammatory Diseases Such As Rheumatoid Disease, Fever And Systemic Infection Which Will Confound The Level Of Serum CRP
* Patients With Known Intolerance, Contraindication Or Hypersensitivity To Losartan, Amlodipine and Hydrochlorothiazide
* Patient With Myocardial Infarction Within The Recent Three Months
* Anatomy Abnormality Which Results In Poor Bilateral Temporal Acoustic Windows Which Prevent TCD Procedure
* Patient Who Requires Continuous Medication With Alpha Blocking Agents
* Concurrent Usage Of Acei
* Poor Mental Function Or Any Other Reason To Expect Difficulty In Meeting The Requirements Of The Study
* Concurrent Treatment With Other Lipid-Lowering Drug
* Childbearing Potential Women Not Undergoing Adequate Contraceptive Control

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-06; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
MCAFV and TCD for measuring cerebral autoregulatory indices at week 0, week 6, week 18 and week 30. | At week 0, week 6, week 18 and week 30.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC